CLINICAL TRIAL: NCT05476692
Title: Clinical Outcome of Surgical Treatment for Osteochondral Lesions of the Talus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Magdy Fahmy Dawood, Principal Investigator, Assiut University
Other Study IDs: OCD of the talus
Record Dates: First submitted 2022-07-18; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Osteochondral Lesion of Talus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AOFAS score and VAS — Clinical outcome by the Visual analogue scale (VAS) and the American Orthopaedic Foot and Ankle (AOFAS) score.

SUMMARY:
Assess clinical and radiological outcome of the various surgical techniques for treatment of osteochondral lesions of the talus

DETAILED DESCRIPTION:
Osteochondritis dissecans (OCD) of the talus is a subchondral bone pathology that presents as an osteochondral lesion of the talar dome with consequent articular cartilage abnormalities. Osteochondral lesions of the talus (OLT) are frequent after acute ankle trauma. The natural history of the OLT remains unclear due to paucity of longitudinal follow-up studies. Various treatment strategies have been described for OLT, including conservative treatment and operative treatment However, the current literature does not allow firm evidence-based recommendations concerning the treatment to be established ; Microfracture is the most common reparative surgery for osteochondral lesions of the talus (OLTs). While shown to be effective in short- to midterm outcomes, the fibrocartilage that microfracture produces is both biomechanically and biologically inferior to that of native hyaline cartilage and is susceptible to possible deterioration over time following repair . Arthroscopic debridement (AD) for the osteochondral lesions of the talar dome (OLT) was widely documented in the nineties with satisfactory results. However, in modern treatment algorithms, its role is not described. A frequently used instrument for assessing outcome after ankle and hindfoot injuries is the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score .

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 60 years old.
* Traumatic and degenerative etiology.
* without ankle deformity.
* No inflammatory arthritis.
* Absent or corrected ligamentous instability

Exclusion Criteria:

* Older than 60 years old and younger than 15 years old.
* Charcot ankle.
* Vascular injury.

Ages: 15 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: the study is a descriptive case series study. The sample will be included from the admitted 40 patients during 12 months from the start of the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
clinical outcome of the various surgical techniques for treatment of osteochondral lesions of the talus | 1 year
  clinical outcome of the various surgical techniques for treatment of osteochondral lesions of the talus , Clinical outcome by the AOFAS score ( American Orthopaedic Foot and Ankle Society), the higher score means the better outcome and the lower score means the worse outcome

REFERENCES:
- See also: Management of Osteochondral Lesions of the Talar Dome — https://pubmed.ncbi.nlm.nih.gov/28979588/
- See also: Osteochondritis dissecans of the talus — https://pubmed.ncbi.nlm.nih.gov/25606554/
- See also: Long-term Outcomes of Microfracture for Treatment of Osteochondral Lesions of the Talus — https://pubmed.ncbi.nlm.nih.gov/33719632/